CLINICAL TRIAL: NCT05977140
Title: A Phase 1, Randomized, Double-Blinded, Placebo-Controlled, First-in-Human Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single-Ascending and Multiple-Ascending Doses of Oral CDI-988 in Healthy Adult Participants
Brief Title: CDI-988 Safety Study in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cocrystal Pharma, Inc. (Industry)
Collaborators: Cocrystal Pharma Australia Pty Ltd. (Unknown); Beyond Drug Development Pty Ltd. (Unknown); Resolutum Global Pty Ltd. (Unknown); Scientia Clinical Research Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDI-988-P1-001
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
Keywords: Coronavirus; SARS-CoV-2
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Part 1: 5 randomized single ascending dose cohorts of 8 participants and 1 open-label single ascending dose cohort of 6 participants. In Part 2, 6 multiple ascending dose cohorts, each with 8 participants
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- SAD Cohort 1A (Experimental): first single-dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- SAD Cohort 1B (Experimental): second single-dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- SAD Cohort 1C (Experimental): third single-dose level; food-effect cohort
  Interventions: Drug: CDI-988; Drug: Placebo
- SAD Cohort 1D (Experimental): fourth single-dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- MAD Cohort 2A (Experimental): first multiple-dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- MAD Cohort 2B (Experimental): second multiple-dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- MAD Cohort 2C (Experimental): third multiple-dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- SAD Cohort 1E (Experimental): fifth dose level; food effect cohort
  Interventions: Drug: CDI-988; Drug: Placebo
- SAD Cohort 1F (Experimental): sixth dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- MAD Cohort 2D (Experimental): 4th multiple dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- MAD Cohort 2E (Experimental): 5th multiple dose level
  Interventions: Drug: CDI-988; Drug: Placebo
- MAD Cohort 2F (Experimental): 6th multiple dose level
  Interventions: Drug: CDI-988; Drug: Placebo

INTERVENTIONS:
Drug: CDI-988 — SARS-CoV-2 3CL protease inhibitor
Drug: Placebo — matching placebo

SUMMARY:
The goal of this clinical trial is to learn about the safety and pharmacokinetics (PK, the amount of drug in the blood) of a new drug called CDI-988 in healthy volunteers.

The main questions it aims to answer are:

* Are there any side effects of the drug?
* What is the amount of drug that reaches the bloodstream? Participants will be assigned by chance to take either CDI-988 or placebo by mouth and have physical exams, electrocardiograms (ECGs), vital signs, and blood tests to look for any side effects.

DETAILED DESCRIPTION:
CDI-988 is a severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) 3-chymotrypsin-like (3CL) protease inhibitor for oral administration. This study is being conducted in 2 parts to examine the safety, tolerability, and PK of CDI-988 in healthy participants. Part 1 will entail escalating single doses in sequential cohorts and Part 2 will enroll escalating multiple-dose cohorts. Participants will be monitored for adverse events, vital signs, laboratory values, and electrocardiograms (ECGs).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or non-pregnant, non-lactating females
* Body weight of at least 45 kg.
* Body mass index ≥18.0 and ≤32.0 kg/m2
* Good state of mental and physical health
* Negative severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) test

Exclusion Criteria:

* Received an investigational drug within 30 days
* Received a coronavirus disease 2019 (COVID-19) vaccine within 7 days
* Drug or alcohol abuse in the past 12 months
* Clinically significant abnormal biochemistry, hematology, coagulation, urinalysis test results
* Clinically significant abnormal ECG or vital signs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2025-05-23 (Actual); Study Completion 2025-07-23 (Actual)

PRIMARY OUTCOMES:
Adverse events | Day 1 to 7 days after last dose
  number of participants with treatment-emergent adverse events
Laboratory abnormalities | Day 1 to 7 days after last dose
  number of participants with clinically significant laboratory abnormalities
Vital signs | Day 1 to 7 days after last dose
  number of participants with clinically significant changes from baseline in vital signs
ECGs | Day 1 to 7 days after last dose
  number of participants with clinically significant changes from baseline in ECGs

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 to 3 days after last dose
Time of maximum plasma concentration (Tmax) | Day 1 to 7 days after last dose
Area under the plasma concentration-time curve (AUC) | Day 1 to 3 days after last dose
Elimination rate constant (lambda Z) | Day 1 to 3 days after last dose
Terminal elimination half-life (t1/2) | Day 1 to 3 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Argent, MD, Principal Investigator — Scientia Clinical Research
Locations (1):
- Scientia Clinical Research Pty Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No